CLINICAL TRIAL: NCT00259467
Title: Tailored Activity to Improve Affect in Dementia
Brief Title: Project TAP: Tailored Activities Project
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Laura N. Gitlin, Ph.D, Jefferson Center for Applied Research on Aging and Health
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: R21MH069425 (NIH)
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Alzheimer's Disease
Keywords: Activity, Dementia, Caregiving
MeSH Terms: conditions — Alzheimer Disease; Motor Activity; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Home-Based Behavorial Intervention

SUMMARY:
Specific Aims

1. Establish a preliminary effect size for the impact of the intervention on depressive affect and agitated behaviors in persons with dementia in 4 months
2. Evaluate acceptance of and engagement in activities in persons with dementia
3. Establish a preliminary effect size for the impact of the intervention on caregiver burden, depressive symptoms, and mastery at 4 months.
4. Evaluate caregiver skills acquisition, acceptance of and compliance to intervention techniques.

ELIGIBILITY:
Inclusion Criteria:

* Care Recipient
* English Speaking
* NINCDS-ADRDA diagnosis[physician generated of dementia or mini-mental state examination score of less than or equal to 23;3] Able to feel self; and participates in at least 2 other activities of daily living[ADLs-Bathing, Dressing, Grooming, Toileting, Transferring from bed to chair] As reported by caregiver.
* Caregiver
* English Speaking
* Family member 21 years of age or older [male or female]
* Lives with Care Recipient
* Has telephone in the home
* Plans to live in area for 8 months
* Indicated willingness to learn new approaches by which to engage care recipient in meaningful activities
* Provides 4 or more hours a day directly caring or providing for care recipient

Exclusion Criteria:

* Care Recipient
* Has Schizophrenia or Bi-Polar Disorder
* Their Dementia is secondary to probable head trauma
* Their MMSE score is equal to zero and they are bed bound, defined as confinement to bed or chair for at least 22 hours a day for at least 4 of 7 days
* They are not responsive to their environment
* Caregiver
* Are currently involved in another clinical trial of psycho-social or educational interventions for caregivers
* Are planning to place their family member in a nursing home within the next 8 months. Also, the care recipient/caregiver dyad will be excluded if either caregiver or care recipient: 1) has a terminal illness with life expectancy less than 8 months 2)is in active treatment for cancer or 3) has had greater than 3 acute medical hospitalizations within the past year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-02; Study Completion 2007-01

PRIMARY OUTCOMES:
Behavioral occurrence
Care recipient depressive mood
Caregiver upset

SECONDARY OUTCOMES:
Activity engagement and vigilance

CONTACTS AND LOCATIONS:
Overall Officials: Laura N Gitlin, Ph.D, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gitlin LN, Winter L, Vause Earland T, Adel Herge E, Chernett NL, Piersol CV, Burke JP. The Tailored Activity Program to reduce behavioral symptoms in individuals with dementia: feasibility, acceptability, and replication potential. Gerontologist. 2009 Jun;49(3):428-39. doi: 10.1093/geront/gnp087. Epub 2009 May 6. PMID 19420314